CLINICAL TRIAL: NCT02099721
Title: Improve Sudden Cardiac Arrest Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Improve SCA
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Sudden Cardiac Arrest; Ventricular Arrythmia
Keywords: Sudden Cardiac Arrest (SCA); Syncope; Non Sustained Ventricular Tachycardia (NSVT); Premature Ventricular Contractions (PVC); Left Ventricular Ejection Fraction (LVEF); Primary Prevention; Secondary Prevention; Antitachycardia pacing (ATP); shock; appropriate therapy
MeSH Terms: conditions — Death, Sudden, Cardiac; Syncope; Ventricular Premature Complexes; Shock | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A: Secondary prevention patients- device implant (Active Comparator): Patients who are guideline indicated for an ICD/CRT-D for secondary prevention of sudden cardiac arrest.
  These subjects receive an ICD/CRT-D implant.
  Interventions: Device: ICD or CRT-D Device
- Group B: Secondary prevention patients - no device implant (No Intervention): Patients who are guideline indicated for an ICD/CRT-D for secondary prevention of sudden cardiac arrest.
  These subjects choose not to receive an ICD/CRT-D implant.
- Group C: 1.5 Prevention patients - device implant (Active Comparator): Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects receive an ICD/CRT-D implant.
  Interventions: Device: ICD or CRT-D Device
- Group D: 1.5 prevention patients - no device implant (No Intervention): Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects choose not to receive an ICD/CRT-D implant.
- Group E: Primary, non-1.5 patients - device implant (Other): Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they do NOT fall into the 1.5 prevention group. These patients do not have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF) which would put them into the 1.5 prevention group.
  These subjects receive an ICD/CRT-D implant.
  Interventions: Device: ICD or CRT-D Device
- Group F: Primary, non-1.5 patients - no device (No Intervention): Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they do NOT fall into the 1.5 prevention group. These patients do not have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF) which would put them into the 1.5 prevention group.
  These subjects choose not to receive an ICD/CRT-D implant.

INTERVENTIONS:
Device: ICD or CRT-D Device — Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming. The programming is not investigational. Consistent programming is desirable in order to compare groups during statistical analysis.
  Arms: Group A: Secondary prevention patients- device implant; Group C: 1.5 Prevention patients - device implant; Group E: Primary, non-1.5 patients - device implant

SUMMARY:
The purpose of this study is to demonstrate that primary prevention patients with one or more additional risk factors (1.5 prevention criteria: syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent pre-ventricular contractions (PVCs), and low left ventricular ejection fraction (LVEF)) are at a similar risk of life-threatening ventricular arrhythmias (LTVA) when compared to secondary prevention patients, and would receive similar benefit from an implantable cardioverter defibrillator (ICD), or cardiac resynchronization therapy- defibrillator (CRT-D) implant.

DETAILED DESCRIPTION:
Devices allowed in the study include any Medtronic single, dual, or triple chamber defibrillator that has received appropriate license or regulatory approval and is commercially available by Medtronic in the geography in which the implant will take place. Any market-released, commercially available lead(s) can be used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Class I indication for implantation of an ICD according to the American College of Cardiology (ACC)/American Heart Association(AHA)/Heart Rhythm Society (HRS) or European Society of Cardiology (ESC) Guidelines
* Subject (or subject's legally authorized representative) is willing and able to sign and date the Patient Informed Consent Form.

Exclusion Criteria:

* Subject is ≤ 18 years of age
* Subject with any exclusion criteria as required by local law (e.g., age, pregnancy, breast feeding)
* Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the Medtronic Clinical Trial Leader
* Subject has any contraindication for ICD/CRT-D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4222 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu Zhang, Principal Investigator — Fuwai Hospital Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (90):
- Argentina (4):
  - Hospital Churruca, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Universitario Fundación Favaloro, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires (ICBA), Buenos Aires
- Republican Scientific and Practical Center "Cardiology", Minsk, Belarus
- Brazil (2):
  - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo, São Paulo
  - INCOR - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo
- China (36):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Xiamen Heart Center, Xiamen, Fujian
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - First Hospital of Dalian Medical University, Dalian, Liaoning
  - The General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Sichuan, Sichuan
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Fuwai Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - The Second Affiliated Hospital of the Third Military Medical University, Chongqing
  - Fujian Provincial Hospital, Fuzhou
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangzhou
  - The First Affiliated Hospital of Sun Yat-Sen Medical University, Guangzhou
  - Guizhou Province People's Hospital, Guiyang
  - The First Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Zhejiang Greentown Cardiovascular Hospital, Hangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Jinhua Municipal Central Hospital, Jinhua
  - Jiangsu Province People's Hospital, Nanjing
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xinhua Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Shenzhen Sun Yat-sen Cardiovascular Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an
- Fundacion Cardioinfantil, Bogotá, Colombia
- Wadi El-Neel Hospital, Cairo, Egypt
- India (13):
  - Care Hospital, Hyderabad, Andhra Pra
  - Medanta- The Medicity, Gurgaon, Haryana
  - Ruby Hall Clinic, Pune, Maharashtr
  - King George's Medical University, Lucknow, Uttar Prad
  - BM Birla Heart Research Centre, Kolkata, West Bengal
  - Care Institute of Medical Sciences (CIMS), Ahmedabad
  - Post Graduate Institute of Medical Education & Research, Chandigarh
  - Lisie Hospital, Kochi
  - B.M. Birla Heart Reserch Centre, Kolkata
  - BM Birla Heart Research CentreB, Kolkata
  - All India Institute of Medical Sciences, New Delhi
  - Govind Ballabh Pant Hospital, New Delhi
  - Krishna Institute of Medical Sciences (KIMS), Secunderabad
- Malaysia (2):
  - Institut Jantung Negara - National Heart Institute, Kuala Lumpur
  - Universiti Malaya Medical Centre, Kuala Lumpur
- Mexico (4):
  - Hospital Angeles Lomas, León, Guanajuato
  - Hospital Angeles Lomas, Huixquilucan de Degollado
  - Hospital Angeles Leon, León
  - Hospital General de Puebla, Puebla City
- Russia (6):
  - Russian Scientific Center of Surgery by B.V. Petrovkiy, RAMN, Moscow
  - Russian Scientific Center of Surgery by B.V. Petrovskiy, RAMN, Moscow
  - Novosibirsk Research Institute of Circulation Pathology, Novosibirsk
  - Scientific Research Institute of Cardiology, Tomsk
  - Tyumen Regional Clinical Hospital, Tyumen
  - Tyumen Cardiology Center, Tyumen
- Singapore (2):
  - Changi General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- Groote Schuur Hospital, Cape Town, South Africa
- South Korea (9):
  - Sejong Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul Saint Mary's Hospital, Seoul
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital Hsin Chu Branch, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Military Hospital, Montfleury, Tunisia
- Dubai Hospital, Dubai, United Arab Emirates

REFERENCES:
- [Derived] Zhao S, Ching CK, Huang D, Liu YB, Rodriguez-Guerrero DA, Hussin A, Kim YH, Van Dorn B, Zhou X, Singh B, Zhang S; Improve SCA Investigators. Regional disparities and risk factors of mortality among patients at high risk of sudden cardiac death in emerging countries: a nonrandomized controlled trial. BMC Med. 2024 Mar 22;22(1):130. doi: 10.1186/s12916-024-03310-5. PMID 38519982
- [Derived] Singh B, Hsieh YC, Liu YB, Lin KH, Joung B, Rodriguez DA, Chasnoits AR, Huang D, Zhang S, O'Brien JE, Lexcen DR, Cerkvenik J, Van Dorn B, Ching CK. Cardioverter-defibrillator reduces mortality risk in eligible ischemic and non-ischemic cardiomyopathy patients: Sub-analysis of the multi-center Improve SCA study. Indian Heart J. 2023 Mar-Apr;75(2):115-121. doi: 10.1016/j.ihj.2023.01.010. Epub 2023 Feb 2. PMID 36736459
- [Derived] Ching CK, Hsieh YC, Liu YB, Rodriguez DA, Kim YH, Joung B, Singh B, Huang D, Hussin A, Chasnoits AR, O'Brien JE, Cerkvenik J, Lexcen D, Van Dorn B, Zhang S. The mortality analysis of primary prevention patients receiving a cardiac resynchronization defibrillator (CRT-D) or implantable cardioverter-defibrillator (ICD) according to guideline indications in the improve SCA study. J Cardiovasc Electrophysiol. 2021 Aug;32(8):2285-2294. doi: 10.1111/jce.15149. Epub 2021 Jul 9. PMID 34216069
- [Derived] Zhang S, Ching CK, Huang D, Liu YB, Rodriguez-Guerrero DA, Hussin A, Kim YH, Chasnoits AR, Cerkvenik J, Lexcen DR, Muckala K, Brown ML, Cheng A, Singh B; Improve SCA Investigators. Utilization of implantable cardioverter-defibrillators for the prevention of sudden cardiac death in emerging countries: Improve SCA clinical trial. Heart Rhythm. 2020 Mar;17(3):468-475. doi: 10.1016/j.hrthm.2019.09.023. Epub 2019 Sep 24. PMID 31561030
- [Derived] Singh B, Zhang S, Ching CK, Huang D, Liu YB, Rodriguez DA, Hussin A, Kim YH, Chasnoits AR, Cerkvenik J, Muckala KA, Cheng A. Improving the utilization of implantable cardioverter defibrillators for sudden cardiac arrest prevention (Improve SCA) in developing countries: Clinical characteristics and reasons for implantation refusal. Pacing Clin Electrophysiol. 2018 Dec;41(12):1619-1626. doi: 10.1111/pace.13526. Epub 2018 Oct 31. PMID 30320410
- [Derived] Zhang S, Singh B, Rodriguez DA, Chasnoits AR, Hussin A, Ching CK, Huang D, Liu YB, Cerkvenik J, Willey S, Kim YH. Improve the prevention of sudden cardiac arrest in emerging countries: the Improve SCA clinical study design. Europace. 2015 Nov;17(11):1720-6. doi: 10.1093/europace/euv103. Epub 2015 Jun 1. PMID 26037794

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Secondary Prevention Patients- Device Implant: Patients who are guideline indicated for an ICD/CRT-D for secondary prevention of sudden cardiac arrest.
  These subjects receive an ICD/CRT-D implant.
  ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming. The programming is not investigational. Consistent programming is desirable in order to compare groups during statistical analysis.
- Group B: Secondary Prevention Patients - no Device Implant: Patients who are guideline indicated for an ICD/CRT-D for secondary prevention of sudden cardiac arrest.
  These subjects chose not to receive an ICD/CRT-D implant.
- Group C: 1.5 Prevention Patients - Device Implant: Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects receive an ICD/CRT-D implant.
  ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming. The programming is not investigational. Consistent programming is desirable in order to compare groups during statistical analysis.
- Group D: 1.5 Prevention Patients - no Device Implant: Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects chose not to receive an ICD/CRT-D implant.
- Group E: Primary, Non-1.5 Patients - Device Implant: Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they do NOT fall into the 1.5 prevention group. These patients do not have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF) which would put them into the 1.5 prevention group.
  These subjects receive an ICD/CRT-D implant.
  ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming. The programming is not investigational. Consistent programming is desirable in order to compare groups during statistical analysis.
- Group F: Primary, Non-1.5 Patients - no Device: Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they do NOT fall into the 1.5 prevention group. These patients do not have one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF) which would put them into the 1.5 prevention group.
  These subjects chose not to receive an ICD/CRT-D implant.
Period: Overall Study
Arm/Group | Group A: Secondary Prevention Patients- Device Implant | Group B: Secondary Prevention Patients - no Device Implant | Group C: 1.5 Prevention Patients - Device Implant | Group D: 1.5 Prevention Patients - no Device Implant | Group E: Primary, Non-1.5 Patients - Device Implant | Group F: Primary, Non-1.5 Patients - no Device
Started | 1066 | 127 | 1068 | 845 | 331 | 452
Completed (Non-exited patients. Patients from China were considered completers if they had a 24 month visit.) | 990 | 0 (Not implanted secondary patients were automatically exited.) | 983 | 774 | 304 | 432
Not Completed | 76 | 127 | 85 | 71 | 27 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Secondary Prevention Patients- Device Implant | Group B: Secondary Prevention Patients - no Device Implant | Group C: 1.5 Prevention Patients - Device Implant | Group D: 1.5 Prevention Patients - no Device Implant | Group E: Primary, Non-1.5 Patients - Device Implant | Group F: Primary, Non-1.5 Patients - no Device | Total
Number analyzed (Participants) | 1066 | 127 | 1068 | 845 | 331 | 452 | 3889
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (14.3) | 55.7 (15.5) | 61.1 (11.7) | 59.1 (13.3) | 61.3 (11.3) | 57.8 (13.7) | 59.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 27 | 253 | 176 | 95 | 103 | 908
  Male | 812 | 100 | 815 | 669 | 236 | 349 | 2981
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One patient in Group F did not specify any of the above categories.
  Participants
    Race / Ethnic Origin: number analyzed (Participants) | 1066 | 127 | 1068 | 845 | 331 | 451 | 3888
    Race / Ethnic Origin: Asian Indian | 159 | 23 | 115 | 273 | 44 | 239 | 853
    Race / Ethnic Origin: Black or African | 7 | 0 | 8 | 2 | 3 | 1 | 21
    Race / Ethnic Origin: Chinese | 529 | 97 | 595 | 475 | 158 | 182 | 2036
    Race / Ethnic Origin: Korean | 229 | 4 | 158 | 25 | 50 | 15 | 481
    Race / Ethnic Origin: Other Asian | 35 | 1 | 28 | 50 | 9 | 5 | 128
    Race / Ethnic Origin: White or Caucasian | 85 | 2 | 119 | 10 | 52 | 4 | 272
    Race / Ethnic Origin: Other Race | 17 | 0 | 42 | 10 | 14 | 5 | 88
    Race / Ethnic Origin: Not reportable per local laws or regulations | 1 | 0 | 1 | 0 | 1 | 0 | 3
    Race / Ethnic Origin: Subject/physician chose not to provide information | 4 | 0 | 2 | 0 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  Colombia | 11 | 0 | 25 | 0 | 6 | 0 | 42
  Argentina | 27 | 0 | 33 | 1 | 21 | 0 | 82
  Singapore | 14 | 5 | 42 | 76 | 23 | 27 | 187
  Egypt | 6 | 2 | 1 | 1 | 1 | 1 | 12
  Malaysia | 45 | 0 | 23 | 30 | 0 | 0 | 98
  United Arab Emirates | 3 | 0 | 3 | 1 | 5 | 0 | 12
  Belarus | 8 | 0 | 7 | 1 | 1 | 0 | 17
  India | 149 | 22 | 104 | 263 | 39 | 236 | 813
  Russia | 21 | 0 | 46 | 0 | 24 | 0 | 91
  South Korea | 232 | 4 | 160 | 25 | 52 | 15 | 488
  China | 385 | 85 | 545 | 359 | 144 | 136 | 1654
  Taiwan | 125 | 9 | 18 | 72 | 1 | 29 | 254
  Brazil | 9 | 0 | 6 | 0 | 0 | 0 | 15
  Mexico | 3 | 0 | 17 | 9 | 5 | 4 | 38
  South Africa | 5 | 0 | 9 | 2 | 3 | 1 | 20
  Tunisia | 22 | 0 | 28 | 5 | 6 | 3 | 64
  Malta | 1 | 0 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Occurrence of a Ventricular Arrhythmia
Description: Time to the first occurrence of an episode of true ventricular tachycardia or fibrillation
  24 Month rates will be provided for the two groups used in the primary endpoint definition. However, the primary endpoint of hazard ratio is presented in Statistical Analysis 1 as a ratio between Groups A and C.
Time Frame: Hazard ratio from study enrollment to approximately 4 years post-implant/enrollment (as reported in Statistical Analysis 1), and estimated 24 month VT-VF rate (as compared in the Outcome Measure table between Groups A and C).
Population: Implanted 1.5 primary prevention and implanted secondary prevention patients. Since the primary objective is the hazard ratio of implanted 1.5 patients to implanted secondary patients, Groups B, D, E and F are not compared for this outcome. While not the primary endpoint, 24-month rates are provided to illustrate the underlying data.
Measure: Number (95% Confidence Interval); unit: Estimated 24-Month VT-VF Pct of Patients
Groups:
- Group A: Secondary Prevention Patients - Device Implant: Patients who are guideline indicated for an ICD/CRT-D for secondary prevention of sudden cardiac arrest.
  These subjects receive an ICD/CRT-D implant.
  ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming. The programming is not investigational. Consistent programming is desirable in order to compare groups during statistical analysis.
- Group C: 1.5 Prevention Patients - Device Implant: Patients who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have any one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects receive an ICD/CRT-D implant.
  ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming. The programming is not investigational. Consistent programming is desirable in order to compare groups during statistical analysis.
Arm/Group | Group A: Secondary Prevention Patients - Device Implant | Group C: 1.5 Prevention Patients - Device Implant
Number analyzed (Participants) | 1053 | 1068
Estimated 24-Month VT-VF Pct of Patients | 32.5 [29.3 to 36.0] | 18.3 [15.6 to 21.5]
Statistical Analysis 1: Comparison: Group A: Secondary Prevention Patients - Device Implant vs Group C: 1.5 Prevention Patients - Device Implant; H0: Hazard ratio of Implanted 1.5 patients (Group C) to implanted secondary patients (Group A) ≤ 0.70 HA: Hazard ratio of Implanted 1.5 patients (Group C) to implanted secondary patients (Group A) > 0.70; Test type: Equivalence — The equivalence margin is a hazard ratio significantly above 0.70; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.38 to 0.57] — The hazard ratio, estimated by a Cox proportional hazard model, has time to first treated VT/VF for 1.5 Prevention in the numerator, with Secondary Prevention in the denominator

2. Secondary Outcome: Mortality
Description: Time to all-cause mortality
Time Frame: Hazard ratio from study enrollment to approximately 4 years post-implant/enrollment (as reported in Statistical Analysis 1), and estimated 24 month mortality rate (as compared in the Outcome Measure table between Groups C and D).
Population: Implanted and not-implanted 1.5 primary prevention patients. Since the secondary objective is the hazard ratio of implanted 1.5 patients to not-implanted 1.5 patients, Groups A, B, E and F are not compared for this outcome. While not the secondary endpoint, 24-month rates are provided to illustrate the underlying data.
Measure: Number (95% Confidence Interval); unit: 24 Mo. Mortality Rate (Pct. of Patients)
Arm/Group | Group C: 1.5 Prevention Patients - Device Implant | Group D: 1.5 Prevention Patients - no Device Implant
Number analyzed (Participants) | 1068 | 845
24 Mo. Mortality Rate (Pct. of Patients) | 12.1 [10.0 to 14.5] | 18.3 [15.6 to 21.5]
Statistical Analysis 1: Comparison: Group C: 1.5 Prevention Patients - Device Implant vs Group D: 1.5 Prevention Patients - no Device Implant; The null hypothesis is that the hazard ratio of implanted to non-implanted 1.5 patients = 1. The alternative is that the ratio is not equal to 1; Test type: Superiority — A hazard ratio significantly below 1 indicates reduced mortality in the 1.5 implanted group; p < 0.0001, Wald chi-square — The p-value is for the effect of treatment group on time to death, adjusting for the baseline covariates of age, gender, QRS duration, ischemic cardiomyopathy, LBBB, NYHA classification, diabetes, LVEF, syncope, NSVT and PVCs; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.40 to 0.66] — Multiple imputations were employed to account for missing baseline covariates

ADVERSE EVENTS:
Time Frame: Baseline through approximately 42 months of follow-up
Description: As the devices in the trial are market approved, adverse event collection was not required to meet study objectives. However, collection of SAEs, serious adverse device events (SADEs) and unanticipated serious adverse device events (USADEs) were mandated in South Korea, Singapore and Taiwan.
  Since only SAEs, SADEs and USADEs in these three countries were collected, Other (Not Including Serious) Adverse Events were not monitored or assessed
Groups:
- Group A: Secondary Prevention Patients - Device Implanted: Patients in South Korea, Singapore and Taiwan who are guideline indicated for an ICD/CRT-D for secondary prevention of sudden cardiac arrest.
  These subjects receive an ICD/CRT-D implant. ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming.
  The programming is not investigational.
  Consistent programming is desirable in order to compare groups during statistical analysis.
- Group B: Secondary Prevention Patients - No Device Implanted: Patients in South Korea, Singapore and Taiwan who are guideline indicated for an ICD/CRT-D for secondary prevention of sudden cardiac arrest.
  These subjects did not receive an ICD/CRT-D implant.
- Group C: 1.5 Prevention Patients - Device Implant: Patients in South Korea, Singapore and Taiwan who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have any one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects receive an ICD/CRT-D implant. ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming.
  The programming is not investigational.
  Consistent programming is desirable in order to compare groups during statistical analysis.
- Group D: 1.5 Prevention Patients - No Device Implant: Patients in South Korea, Singapore and Taiwan who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have any one of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects did not receive an ICD/CRT-D implant.
- Group E: 1.0 Prevention Patients - Device Implant: Patients in South Korea, Singapore and Taiwan who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have none of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects receive an ICD/CRT-D implant. ICD or CRT-D Device: Subjects who receive an ICD/CRT-D device implant will be implanted and follow protocol-specified programming.
  The programming is not investigational.
  Consistent programming is desirable in order to compare groups during statistical analysis.
- Group F: 1.0 Prevention Patients - No Device Implant: Patients in South Korea, Singapore and Taiwan who are guideline indicated for an ICD/CRT-D for primary prevention of sudden cardiac arrest fall into this group if they have none of the 4 additional risk factors (syncope/pre-syncope, non-sustained ventricular tachycardia (NSVT), frequent preventricular contractions (PVCs), or low left ventricular ejection fraction (low LVEF).
  These subjects did not receive an ICD/CRT-D implant.
Arm/Group | Group A: Secondary Prevention Patients - Device Implanted | Group B: Secondary Prevention Patients - No Device Implanted | Group C: 1.5 Prevention Patients - Device Implant | Group D: 1.5 Prevention Patients - No Device Implant | Group E: 1.0 Prevention Patients - Device Implant | Group F: 1.0 Prevention Patients - No Device Implant
All-Cause Mortality (participants affected / at risk) | 33/371 | 0/18 | 24/220 | 24/173 | 3/76 | 4/71
Serious Adverse Events (participants affected / at risk) | 88/371 | 0/18 | 72/220 | 37/173 | 20/76 | 10/71
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Secondary Prevention Patients - Device Implanted (N=371) | Group B: Secondary Prevention Patients - No Device Implanted (N=18) | Group C: 1.5 Prevention Patients - Device Implant (N=220) | Group D: 1.5 Prevention Patients - No Device Implant (N=173) | Group E: 1.0 Prevention Patients - Device Implant (N=76) | Group F: 1.0 Prevention Patients - No Device Implant (N=71)
Cardiac Failure (Cardiac disorders) | 8 (8) | 0 (0) | 21 (30) | 2 (3) | 5 (5) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 3 (3) | 0 (0) | 17 (20) | 1 (1) | 4 (5) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 17 (21) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 6 (7) | 0 (0) | 5 (7) | 3 (8) | 3 (4) | 2 (2)
Pneumonia (Infections and infestations) | 5 (8) | 0 (0) | 4 (4) | 5 (5) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lead dislodgment (Product Issues) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brachiocephalic vein stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brugada syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device lead issue (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device pacing issue (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dystrophic calcification (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart transplant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired hearing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular cyst (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device change (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurogenic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea faciei (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The IMPROVE SCA trial was an non-blinded post-market trial that was not randomized. Thus baseline variables will differ across the treatment groups. Covariate adjustments were made in the analyses as a result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT02099721/SAP_000.pdf
  • Study Protocol (2013-12-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT02099721/Prot_001.pdf